CLINICAL TRIAL: NCT00802568
Title: Pilot Study of Allogeneic Hematopoietic Stem Cell Transplantation Following Reduced Intensity Conditioning in Treating Patients With Multiple Myeloma
Brief Title: Fludarabine, Busulfan, Antithymocyte Globulin, and Donor Stem Cell Transplant in Treating Patients With Multiple Myeloma That Has Not Responded to Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626720; IPC-2005-002; IPC-ITT 04-02; EUDRACT-2005-01053-13; INCA-RECF0428; AMGEN-IPC-2005-002; JANSSEN-IPC-2005-002
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2008-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; osteolytic lesions of multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Antilymphocyte Serum; Busulfan; fludarabine phosphate

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: fludarabine phosphate
Procedure: allogeneic bone marrow transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase II trial is studying the side effects of giving fludarabine together with busulfan and antithymocyte globulin followed by donor stem cell transplant and to see how well it works in treating patients with multiple myeloma that has not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To study the toxicity of reduced intensity conditioning comprising fludarabine phosphate, busulfan, and anti-thymocyte globulin followed by allogeneic hematopoietic stem cell transplantation in patients with refractory or relapsed multiple myeloma.

Secondary

* To study the tumor response in these patients.
* To study the incidence of acute or chronic graft-versus-host disease in these patients.
* To study the incidence of infectious complications in these patients.
* To study relapse- or progression-free and overall survival of these patients.
* To study the biological mechanisms (i.e., taking graft, immunological recovery, antitumor activity, and chimerism).

OUTLINE: This is a multicenter study.

Patients receive reduced intensity conditioning comprising fludarabine IV on days -5 to -1, oral busulfan on days -4 and -3, and anti-thymocyte globulin IV on days -2 and -1. Patients undergo allogeneic hematopoietic stem cell transplantation on day 0.

After completion of study therapy, patients are followed every month for 6 months and then every 3 months for 1½ years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma, meeting 1 of the following criteria:

  * Stage I disease with a bone lesion
  * Stage II or III disease meeting any of the following criteria:

    * Elevated beta-2 microglobulin
    * Deletion of chromosome 13
* Refractory or relapsed disease
* Presence of an evaluable monoclonal component
* Must have achieved reduction of primary tumor after receiving prior intensified chemotherapy with high-dose melphalan and cyclosporine with autologous transplantation
* HLA identical family donor available

  * Bone marrow transplantation is allowed in case hematopoietic stem cell collection fails

PATIENT CHARACTERISTICS:

* Karnofsky 70-100%
* No contraindications to allogeneic transplantation
* No contraindications to drugs used in conditioning regimen
* No psychiatric illness
* No other cancer within the past 5 years except basal cell skin cancer or epithelioma in situ of the cervix
* No serious and uncontrolled infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 1 month since participation in another prior clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mortality rate at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Didier Blaise, MD — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France